CLINICAL TRIAL: NCT06015035
Title: A Prospective Single-center, Single-arm, Open-label Study of Sintilimab and Anlotinib Combined With Chemotherapy in Neoadjuvant Treatment of Resectable Esophageal Cancer
Brief Title: Sintilimab and Anlotinib Combined With Chemotherapy in Neoadjuvant Treatment of Resectable Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Xiaolong Yan, Dr., Deputy director, Tang-Du Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: k202204-02
Record Dates: First submitted 2023-08-17; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Sintilimab and Anlotinib in Combination With Chemotherapy
Keywords: esophageal cancer; neoadjuvant; efficiency
MeSH Terms: conditions — Esophageal Neoplasms | interventions — sintilimab; anlotinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anlotinib for anti-angiogenesis and sintilimab and chemotherapy (Experimental): Neoadjuvant treatment involved administering anlotinib (10 mg orally, once a day, 2 weeks on and 1 week off) for anti-angiogenesis and sintilimab (200 mg) and chemotherapyfor three cycles.
  Interventions: Drug: Sintilimab and anlotinib in combination with chemotherapy

INTERVENTIONS:
Drug: Sintilimab and anlotinib in combination with chemotherapy — Neoadjuvant treatment involved administering anlotinib (10 mg orally, once a day, 2 weeks on and 1 week off) for anti-angiogenesis and sintilimab (200 mg) and chemotherapyfor three cycles. Surgical treatment was performed 4-6 weeks after the last chemotherapy cycle was completed. The primary endpoints assessed were pathological complete response (pCR) rate and safety.

SUMMARY:
The study focused on patients with T2-4NxM0 resectable esophageal carcinoma. Neoadjuvant treatment involved administering anlotinib (10 mg orally, once a day, 2 weeks on and 1 week off) for anti-angiogenesis and sintilimab (200 mg) and chemotherapyfor three cycles. Surgical treatment was performed 4-6 weeks after the last chemotherapy cycle was completed. The primary endpoints assessed were pathological complete response (pCR) rate and safety.

DETAILED DESCRIPTION:
The study was conducted from April 2021 to April 2022 at our hospital and was approved by the Ethics Committee of Tangdu Hospital. The inclusion criteria were as follows: patients aged 18-75 years with a histopathologic diagnosis of esophageal cancer staged according to the AJCC eighth edition as T1-4N1-3M0. If patients were staged as T2N0M0, the esophageal lesions had to be ≥5 cm. Before enrollment, all patients underwent various examinations, including cardiac color ultrasound (left ventricular ejection fraction of at least 50%), pulmonary function (forced expiratory volume-1 [FEV1] ≥1.5 L), enhanced chest computed tomography (CT), abdominal color ultrasound, cervical lymph node color ultrasound and other necessary laboratory tests (such as blood routine, liver and kidney function, electrolytes, and cortisol rhythm) to exclude treatment and surgical contraindications and ensure suitability for ICIs treatment.

The exclusion criteria were as follows: Patients unable to tolerate surgery, those with refractory hypertension and proteinuria, those who had previously received other treatments, and those who were not suitable candidates for ICIs (due to conditions such as hepatitis B with viral quantification >2000 IU, systemic lupus erythematosus, and xerosis).

Treatment regimen:

Patients were administered preoperatively with sintilimab (200 mg, Day 1) and anlotinib (10 mg, orally, once daily, 2 weeks on and 1 week off) in combination with chemotherapy (albumin paclitaxel 130 mg/m2, Days 1 and 8 + nedaplatin 80 mg/m2, Day 1) for three cycles of neoadjuvant therapy. Surgical intervention (either Mckeown or Ivor Lewis approach) was performed 4-6 weeks after completing the last treatment cycle of neoadjuvant therapy. After the 4th week after surgery, patients received maintenance therapy with sintilimab (200 mg, Q3W) for 1 year. If any adverse reactions of grade 3 or higher occurred during the treatment, the dose of chemotherapeutic drugs was reduced by 25% until the patient's condition recovered to grade 1 or returned to normal, and the subsequent treatment cycle was continued. In case of grade 3 or higher hypertension or proteinuria, the dose of anlotinib was reduced to 8 mg. It was discontinued if the condition could not recover to grade 1-2 after symptomatic treatment.

ELIGIBILITY:
Inclusion Criteria

* patients aged 18-75 years with a histopathologic diagnosis of esophageal cancer staged according to the AJCC eighth edition as T1-4N1-3M0. If patients were staged as T2N0M0, the esophageal lesions had to be ≥5 cm.
* Before enrollment, all patients underwent various examinations, including cardiac color ultrasound (left ventricular ejection fraction of at least 50%), pulmonary function (forced expiratory volume-1 [FEV1] ≥1.5 L), enhanced chest computed tomography (CT), abdominal color ultrasound, cervical lymph node color ultrasound ▪ other necessary laboratory tests (such as blood routine, liver and kidney function, electrolytes, and cortisol rhythm) to exclude treatment and surgical ontraindications and ensure suitability for ICIs treatment.

Exclusion Criteria:

* Patients unable to tolerate surgery
* those with refractory hypertension and proteinuria
* those who had previously received other treatments
* those who were not suitable candidates for ICIs (due to conditions such as hepatitis B with viral quantification >2000 IU, systemic lupus erythematosus, and xerosis).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Primary Endpoints: pCR | up to 24 months
  PCR: This was assessed by examining the postoperative pathological tissue for the absence of tumor cells in the primary tumor and lymph nodes.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Hongtao Duan, Xi’an, Shanxi
  - Tangdu Hospital, the Air Force Military University, Xi'an

IPD SHARING:
Plan to Share IPD: Undecided
If the clinical study obtains positive results, it will further expand the study